CLINICAL TRIAL: NCT00161213
Title: Phase II Study of Imatinib Mesylate and Gemcitabine for First-line Treatment of Metastatic Pancreatic Cancer
Brief Title: Gemcitabine and Imatinib Mesylate as First-Line Therapy in Patients With Locally Adv. or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000539409; P30CA072720 (NIH); CINJ-070501 (Other: CINJ); CINJ-5324 (Other: CINJ); CINJ-NJ1205 (Other: CINJ)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and Imatinib (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: imatinib mesylate

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine together with imatinib mesylate may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with imatinib mesylate works as first-line therapy in treating patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the time to progression in patients with locally advanced or metastatic pancreatic cancer treated with gemcitabine hydrochloride and imatinib mesylate as first-line therapy.

Secondary

* Assess the response rate in patients treated with this regimen.
* Assess the percentage of patients treated with this regimen who survive 1 year or more.
* Assess the toxicity of this regimen in these patients.
* Assess the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, nonrandomized, open-label, uncontrolled study.

Patients receive gemcitabine hydrochloride IV over 120 minutes on days 3 and 10 and oral imatinib mesylate on days 1-5 and 8-12. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma or poorly differentiated carcinoma (originating in the pancreas)

  * Locally advanced or metastatic disease
* Not eligible for curative resection
* Must have measurable or evaluable disease as defined by RECIST criteria

  * No CA19-9 elevation as only evidence of disease
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 125,000/mm³
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase < 3 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No coexisting medical condition that would preclude study compliance
* No inability to ingest tablets
* No active illness (e.g., active or uncontrolled infection, uncontrolled cardiac disease) that would preclude study participation
* No chronic uncontrolled diarrhea and/or daily emesis
* No other cancer within the past 5 years except for surgically removed noninvasive nonmelanoma skin cancer or in situ cervical cancer

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease
* No prior gemcitabine
* No prior imatinib mesylate
* Prior surgical resection and adjuvant fluorouracil chemotherapy allowed provided there was an interval of > 6 months between the last dose of adjuvant chemotherapy and recurrence of pancreatic cancer
* Prior fluorouracil as a radiosensitizing agent allowed
* At least 4 weeks since prior radiotherapy and recovered

  * Must have evidence of disease outside the radiation fields OR radiologically confirmed disease progression within the radiation fields after completion of radiotherapy
* No concurrent therapeutic warfarin

  * Prophylactic warfarin ≤ 1 mg daily allowed for prophylaxis of central venous catheter thrombosis
  * Low molecular weight heparin or heparin allowed for anticoagulation
* No concurrent chronic systemic corticosteroids
* No other concurrent agents or therapies, including chemotherapy, immunotherapy, hormonal cancer therapy, radiotherapy, or cancer surgery
* No other concurrent experimental medications
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Poplin, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (8):
- United States (8):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CentraState Medical Center, Freehold, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Central Jersey Oncology Group, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - New Jersey Medical School, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moss RA, Moore D, Mulcahy MF, Nahum K, Saraiya B, Eddy S, Kleber M, Poplin EA. A Multi-institutional Phase 2 Study of Imatinib Mesylate and Gemcitabine for First-Line Treatment of Advanced Pancreatic Cancer. Gastrointest Cancer Res. 2012 May;5(3):77-83. PMID 22888387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period spanned from October 2005 through July 2009. The trial was opened at a single regional cancer center and then expanded to other centers to reach accrual goals within the target period. These included hospitals in the CINJ Oncology Group and Northwestern University's Robert H. Lurie Comprehensive Cancer Center.
Groups:
- Gemcitabine and Imatinib: imatinib mesylate: 400 mg/day, given orally Day 1-5 and 8-12 every 21 days.
  gemcitabine hydrochloride: fixed dose rate infuration at 1200 mg/m2/120 minutes on Days 3 and 10 every 21 days.
Period: Overall Study
Arm/Group | Gemcitabine and Imatinib
Started | 44
Completed | 42
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Evaluable for toxicity but not response | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Imatinib
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival in months. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 4 years
Population: A total of 44 patients were enrolled. One patient withdrew consent before starting treatment. One patient was determined, after initiating treatment, to have an ampullary cancer and was evaluable for toxicity but not for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Imatinib
Number analyzed (Participants) | 42
months | 3.9 [2.06 to 5.14]

2. Secondary Outcome: Response Rate
Description: Response rate as defined by a best response of "Stable Disease or better."
Time Frame: 5 years
Population: A total of 44 patients were enrolled. One patient withdrew consent before starting treatment. One patient was determined, after initiating treatment, to have an ampullary cancer and was evaluable for toxicity but not for response. Seven subjects were not assessed for response as they discontinued therapy treatment before response was assessed.
Measure: Number (95% Confidence Interval); unit: percentage of total evaluable subjects
Arm/Group | Gemcitabine and Imatinib
Number analyzed (Participants) | 35
percentage of total evaluable subjects | 48.6 [33.0 to 64.4]

3. Secondary Outcome: 1-year Survival Rate
Description: Percentage of subjects who survive up to 1 year
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of total evaluable subjects
Arm/Group | Gemcitabine and Imatinib
Number analyzed (Participants) | 42
percentage of total evaluable subjects | 25.6 [13.8 to 39.1]

4. Secondary Outcome: Overall Survival
Time Frame: 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Imatinib
Number analyzed (Participants) | 42
months | 6.23 [5.15 to 8.46]

ADVERSE EVENTS:
Time Frame: 5 years
Description: All patients who received one dose of protocol therapy were evaluated for toxicity.
Arm/Group | Gemcitabine and Imatinib
Serious Adverse Events (participants affected / at risk) | 6/43
Other Adverse Events (participants affected / at risk) | 39/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Imatinib (N=43)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (3)
Pain - Abdomen not otherwise specified (Gastrointestinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/thrombus/embolism - pulmonary embolus (Vascular disorders) | 1 (1)
Mood alteration - Depression - pre-existing condition (Psychiatric disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Biliary tree (Infections and infestations) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage, GI - Lower GI NOS (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 (1)
Stricture/stenosis (including anastomotic), GI - Biliary tree (Gastrointestinal disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Imatinib (N=43)
Nausea (Gastrointestinal disorders) | 22 (97)
Constipation (Gastrointestinal disorders) | 12 (15)
Anorexia (Gastrointestinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 9 (9)
Dehydration (Gastrointestinal disorders) | 4 (4)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 25 (66)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 20 (42)
Hemoglobin (Blood and lymphatic system disorders) | 17 (31)
Platelets (Blood and lymphatic system disorders) | 12 (30)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 19 (27)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 9 (11)
Weight loss (General disorders) | 5 (5)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (4)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (3)
Pain - Abdomen NOS (General disorders) | 11 (18)
Pain - Back (General disorders) | 3 (3)
Pain - Other (Specify, __) (General disorders) | 3 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (6)
Memory impairment (Nervous system disorders) | 4 (4)
Confusion (Nervous system disorders) | 3 (3)
Mood alteration - Depression (Psychiatric disorders) | 3 (3)
Edema: limb (Blood and lymphatic system disorders) | 8 (9)
Thrombosis/thrombus/embolism (Vascular disorders) | 5 (8)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes